CLINICAL TRIAL: NCT02605538
Title: Hepatitis B in Cystic Fibrosis and Latent Tuberculosis Respectively
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Time and resource deficiency at the Stockholm CF Center.
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ferenc Karpati, MD, MD, PhD, Karolinska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012/251-31/2
Record Dates: First submitted 2015-05-04; First posted 2015-11-16 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis; Hepatitis A; Hepatitis B; Tuberculosis
MeSH Terms: conditions — Cystic Fibrosis; Hepatitis A; Hepatitis B; Tuberculosis | interventions — Vaccination; twinrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystic Fibrosis (Active Comparator): Vaccination with Twinrix (TM), 3 doses within 6 months according to the manufacturer's instruction. The response will be studied in a time frame of 6 months.
  Interventions: Biological: Vaccination with vaccine against hepatitis A and B
- Healthy volunteers (Active Comparator): Vaccination with Twinrix (TM), 3 doses within 6 months according to the manufacturer's instruction. The response will be studied in a time frame of 6 months.
  Interventions: Biological: Vaccination with vaccine against hepatitis A and B

INTERVENTIONS:
Biological: Vaccination with vaccine against hepatitis A and B — Vaccination against hepatitis A and B
  Other Names: Twinrix (TM)

SUMMARY:
CF patients are at risk for hepatic disease. Vaccination is recommended to all CF patients according to European consensus. The aim of the study is to vaccinate as many patients as possible and to follow up whether immunization has been complete.

DETAILED DESCRIPTION:
Initially, healthy volunteers will be vaccinated to be compared with patients' antibody response to hepatitis A and B vaccine.

The connected part of this study is to vaccinate children suffering from latent tuberculosis against hepatitis B and to measure whether the immunization is related to specific interferon gamma response against Mycobacterium tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* CF patients not previously immunized against hepatitis A or B
* Healthy volunteers not previously immunized against hepatitis A or B
* Age over 1 year

Exclusion Criteria:

* Previously transplanted patients
* Previous vaccination with hepatitis vaccine
* Known allergy against components in Twinrix (TM)

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive antibody response to vaccination with Twinrix(TM) in CF patients compared to healthy volunteers | 6 months for vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ferenc Karpati, MD, PhD, Principal Investigator — Stockholm CF Center, Karolinska University Hospital
Locations (1):
- Stockholm CF Center, KArolinska University Hospital, Stockholm, Sweden